CLINICAL TRIAL: NCT05621785
Title: The Effect of Postnatal Corticosteroid Use on Lung Ultrasonography Scores in Preventing the Development of Bronchopulmonary Dysplasia in Premature Infants
Brief Title: Corticosteroid Use in Premature Babies and Lung Ultrasonografi Use in the Progression to Bronchopulmonary Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sevde Nur Vural, Asistant Doctor, Kırıkkale University
Other Study IDs: Kırıkkale University Faculty
Record Dates: First submitted 2022-11-04; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Bronchopulmonary Dysplasia; Premature Birth
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

INTERVENTIONS:
Device: Lung Ultrasonografi — All babies under 32 weeks of gestation will be included in the study. All data of postnatal corticosteroid users will be recorded using lung USG
  Other Names: corticosteroid

SUMMARY:
Bronchopulmonary dysplasia (BPD) is one of the most common morbidities in premature infants and is associated with poor neurodevelopmental outcomes . Although mechanical ventilation and oxygen requirements in premature infants have been identified as triggering mechanisms for the development of inflammation and BPD over time, data now support that a number of perinatal events that may stimulate the inflammatory cascade before birth also have important effects. Corticosteroids such as dexamethasone and hydrocortisone have proven to be beneficial for the prevention and management of postpartum BPD due to their anti-inflammatory properties . With this study, the effects of corticosteroid use on lung ultrasound findings in BPD will be investigated, and acute and chronic lung ultrasonography scores will be recorded. A prospective observational study was planned in the neonatal intensive care unit between 2022 and 2024 in premature infants below 32 weeks of gestational age. Demographic data and Lung Ultrasonography findings of these babies will be recorded. Among the patients who are predicted to go to BPD, in the group using corticosteroids, Lung Ultrasonographic imaging will be performed and the effect of corticosteroids on pulmonary findings will be recorded. It is planned to investigate whether postnatal steroid use has an effect on lung ultrasound findings in preterm infants with BPD.

DETAILED DESCRIPTION:
It is aimed to show the changes in lung ultrasound findings before, during and after steroid use in premature newborn babies born under 32/7 weeks. Thus, detailed new information will be obtained about the role and importance of corticosteroids in preventing the progression to BPD.

Postnatal corticosteroids are not routinely used to prevent BPD in our unit in our hospital. However, if premature babies meet the following criteria, postnatal low-dose corticosteroids are administered.

In the postnatal third week;

1. Premature infants who are still not weaned from invasive mechanical ventilation.
2. Those who continue to need non-invasive positive pressure ventilation
3. Those who need more than 50% oxygen

Applied steroid protocols:

Dexomethasone:

Total cumulative dose 0.89 mg/kg

* 0.075 mg/kg/dose PO/IV (every 12 hours) for 3 days
* 0.05 mg/kg/dose PO/IV (every 12 hours) 3 days
* 0.025 mg/kg/dose PO/IV (every 12 hours) 2 days
* 0.01 mg/kg/dose PO/IV (every 12 hours) 2 days

Hydrocortisone:

* 1 mg/kg/dose IV/PO (every 12 hours) 7 days
* 0.5 mg/kg/dose IV/PO (every 12 hours) 3 days

Dexsometasone treatment is given in accordance with the DART protocol in infants who cannot wean from invasive mechanical ventilation in accordance with the protocols in use in our unit, which corticosteroid will be used. . In clinical follow-up, corticosteroid preference can be changed by the consultant neonatal specialist according to the general clinical condition of the patient and the accompanying spectrum. Which corticosteroid will be preferred in this observational study will not be known by the team that will conduct the study and will be recorded later.

If more than one corticosteroid use is required in the follow-up, pulmonary ultrasonography findings during the first corticosteroid use will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Those who were born in Kırıkkale University Faculty of Medicine Hospital or who were born in other hospitals and were admitted to Kırıkkale University Faculty of Medicine Neonatal Intensive Care Unit within the first 48 hours of life.
2. Gestational age below 32/7 weeks
3. Those who will be administered postnatal corticosteroids with the decision of the consultant by meeting the diagnostic criteria for going to BPD
4. Informed consent was obtained from the family

Exclusion Criteria:

1. Those with cyanotic congenital heart disease
2. Those with lung and thorax malformations,
3. Those with major congenital anomalies
4. Newborns who do not meet the criteria for postnatal corticosteroid therapy or who are not given postnatal corticosteroids by the consultant
5. The family's refusal to give informed consent

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Gestational age below 32/7 weeks, both sex premature infants
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Bronkopulmoner Displazi under the corticosteroid | 2 years
  Although the use of corticosteroids in the course of BPD has a positive effect on lung ultrasound findings in the acute period in premature newborn babies, long-term beneficial effects cannot be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Sevde Nur Vural, Asistant Dr, Principal Investigator — KIRIKKALE UNİVERSİTY FACULTY OF MEDİCİNE
Locations (1):
- Kırıkkale University Faculty of Medicine, Kırıkkale, Turkey (Türkiye)

REFERENCES:
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896